CLINICAL TRIAL: NCT02749266
Title: The Impact of Chiropractic Activator Adjustments on Mental Rotation and Line Judgment Reaction Time: A Pilot Study
Brief Title: The Impact of Chiropractic Activator Adjustments on Mental Rotation and Line Judgment Reaction Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I-0011
Record Dates: First submitted 2014-07-18; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Cognition - Other
Keywords: chiropractic, cognition
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chiropractic Activator Adjustment (Experimental): Participant will receive a chiropractic adjustment utilizing a handheld chiropractic instrument called an Activator.
  Interventions: Other: Chiropractic adjustment
- Chiropractic sham adjustment (Sham Comparator): Participant will receive a sham (simulated) chiropractic adjustment utilizing a handheld chiropractic instrument called an Activator.
  Interventions: Other: Sham chiropractic adjustment

INTERVENTIONS:
Other: Chiropractic adjustment — Participant will receive a chiropractic adjustment utilizing a handheld chiropractic instrument called an Activator.
  Other Names: Chiropractic Activator adjustment; Chiropractic manipulation
  Arms: Chiropractic Activator Adjustment
Other: Sham chiropractic adjustment — Participants will receive a simulated chiropractic adjustment with a handheld adjusting instrument called an Activator.
  Other Names: Sham manipulation
  Arms: Chiropractic sham adjustment

SUMMARY:
The purpose of this pilot study will be to assess the impact of chiropractic Activator adjustments on spatial cognitive abilities through initial assessment and testing in a healthy population aged 18 to 35.

DETAILED DESCRIPTION:
This study seeks to assess the impact of chiropractic on cognition. Participants must be between 18 and 35 years of age. Within the past six months individuals may not participate if they have had any broken bones, accidents, or surgeries to their spine. Additionally, participants cannot have any mental disabilities, be pregnant, or have other conditions of the spine such as bone mineral loss.

Patients will receive a chiropractic exam and will be randomized to a sham (simulated chiropractic adjustment) or chiropractic adjustment intervention group. Prior to receiving either the sham or chiropractic adjustment, the participants will sit in front of a computer screen and will be asked to follow instructions and press a button on a keypad. There will be three different types of computer assessments that will take approximately fifteen minutes total. After the computer assessments the participant will receive either the sham or chiropractic adjustment. The chiropractic adjustment and the sham will both utilize a handheld instrument called an Activator. After the adjustment or sham the participant will take the computer assessments again. The total time this may take is ninety minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35
* In good health

Exclusion Criteria:

* pregnant
* medically diagnosed cognitive deficits
* medically diagnosed learning disabilities
* fractures, traumas, or surgeries to the spine within the past six months
* diagnosed osteoporosis, articular instability

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Reaction time | Pre and Post intervention (average of 90 minutes)
  Reaction time assessment of keyboard responses to computerized stimulus presentations

SECONDARY OUTCOMES:
Response correctness | Pre and post intervention (average of 90 minutes)
  Correct response to computerized stimulus presentations

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, D.C., Principal Investigator — Life University
Locations (1):
- Life University, Marietta, Georgia, United States